CLINICAL TRIAL: NCT05458882
Title: Impact of an Educational Tool on Quality of Life and Anxiety in Parents of Young Children With Newly Diagnosed Nut Allergy
Brief Title: Impact of an Educational Tool on Quality of Life and Anxiety in Parents of Children With Nut Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health Ireland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 120420
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Child Allergy; Food Allergy
Keywords: Educational intervention; Food allergy; Quality of Life; Anxiety; Self efficacy; Maternal education; Booklet
MeSH Terms: conditions — Food Hypersensitivity; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- educational Booklet (Experimental): Receive intervention- educational booklet describing the day to day social activities and eating out habits of children with established food allergy in Ireland
  Interventions: Behavioral: "living with food allergy" educational booklet
- Routine education (Active Comparator): This group will receive routine education in the allergy group.
  Interventions: Behavioral: "living with food allergy" educational booklet

INTERVENTIONS:
Behavioral: "living with food allergy" educational booklet — An educational booklet giving information on social and eating out habits as well as reaction rates in food allergy Irish children.

SUMMARY:
The number of young children with food allergy, in particular with nut allergy, is increasing worldwide. A diagnosis of nut allergy can cause much anxiety in parents. They worry about their child being exposed to nuts in foods when outside the home. This anxiety can lead to these young children being restricted from taking part in normal childhood activities.

Last year, the investigators conducted a study Recording accidental allergic reactions in children's and teenagers (ReAACT) in which they surveyed over 500 children with food allergy attending our clinic, in order to learn more about their participation in social activities and their practices in relation to eating outside the home.

In the present study, the investigators wish to build upon these results through using the findings to develop a programme to help to lessen the fear and anxiety experienced by parents of young children with newly diagnosed nut allergy. The investigators imagine that knowledge of how other families with children who have food allergy participate in activities involving food outside of the home might help newly diagnosed families.

The investigators would like to know if parents of young children newly diagnosed with nut allergy would benefit from hearing this information. In order to do this, the investigators have developed a short online programme that parents can take part in, in their own homes. Content will focus on the day to day social activities of children with food allergy, based on the findings of the REAACT study. To help the investigators to measure the effectiveness of this programme on reducing anxiety and improving quality of life, they are asking all volunteer participants to complete 4 questionnaires. Two of these questionnaires will ask a parent to indicate 1) the impact of their child's nut allergy on their quality of life and 2) on their child's quality of life. The third questionnaire will ask about their level of anxiety. The fourth questionnaire will ask about their emotions and the coping strategies they use in the context of their child's food allergy.

Participants will be randomized into 2 groups. Group 1 will take part in the online education session along with the usual education provided by the allergy team. The questionnaires will be completed online using only a study identifier number. This will ensure anonymity throughout the study. The only personal information that will be asked is parent's age group, whether they are a mother or father, their child's age and gender and whether they have any other allergies.

Two weeks following the online educational session, Groups 1 and 2 will again complete the online questionnaires.

The research question is to determine if the online educational session is effective at decreasing anxiety and improving quality of life in parents of young children with nut allergy. The outcomes are health related quality of life and level of anxiety. It is hoped that the findings will positively support parents, children and their families in Ireland who are living and managing nut allergy on a daily basis.

DETAILED DESCRIPTION:
Over 4% of children in Ireland have a food allergy. Many studies report that parents and children with food allergy have a decreased quality of life (QOL). However maternal anxiety and parental overprotection even in the absence of FA can lead to childhood anxiety. Children with FA are at risk of exclusion from social activities and overly restrictive lifestyles as parents attempt to minimise risk and their own anxiety by avoiding food related activities. The investigator's department carried out a prospective observation study collecting data on lifestyle practice of food allergic children between 2-16 years attending their services and the rate of accidental allergic reactions (AARs) over 1 year (Recording accidental allergic reactions in children with food allergy: REAACT).

Most children in REACCT (which represents 25% of the return waiting list population) are attending social activities and visiting food venues.

Caregivers can be influenced by high profile media cases which often report fatal AARs occurring in food establishments and during social activities such as parties. The psychological theories of availability heuristic (people make judgements on the likelihood of an event on how easily a case comes to mind) and base case neglect (erroneously judge the likelihood of a situation by failing to consider all relevant data, instead, focusing on new information) can help explain how heavy reporting of rare severe/fatal AAR cases in the media can increase anxiety among vulnerable parents and children leading to social exclusion and avoidance of visiting eateries.

Conversely, there is no reporting of the thousands of food allergic children and families who successfully manage their food allergies and manage to navigate events such as eating out and social activities where food is an integral part. Hence, it is likely that families newly diagnosed with nut allergy are not aware of how other families with established nut allergy behave on a day to day basis.

A primary goal of the allergy clinic is to promote safe, age appropriate, social interaction and eating out behaviors. Therefore, the investigators are interested in finding out whether awareness of the successful management by a greater number of families with nut allergy in Ireland, would impact on level of anxiety and health related quality of life of those newly diagnosed with nut allergy? The investigators hypothesize that providing newly diagnosed children and their parents with information on how other Irish children with established food allergies behave in situations involving food will have a positive impact on their quality of life and level of anxiety and promote "living with risk" rather than "living with fear".

Specifically, they aim to assess the effectiveness of a psycho-educational intervention (illustrating the routine practices of food allergic children regarding social activities and eating out) on disease-speciﬁc quality of life and level of anxiety of newly diagnosed parents and children.

A randomized control trial will be performed comparing quality of life, anxiety and self efficacy in parents who receive the intervention versus those that do not. These parents will have a young child with a newly diagnosed nut allergy.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children between 6 and 36 months
* Parent of children with a new diagnosis of a nut allergy defined as a clinical reaction with a skin prick test (SPT) of >3mm or sensitised with a SPT of >7mm.

Exclusion Criteria:

* Parents who already had a child with a food allergy as parents would have well established coping mechanisms
* Participation in another research project
* Their food allergic child had another chronic condition that might cause anxieties in social environments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1 | 4 weeks
  Change in score in each group on Food allergy Quality of Life Questionnaire (FAQLQ) parental proxy form
Primary Outcome 2 | 4 weeks
  Change in score in each group on Food Allergy Quality of Life (FAQOL) parental burden form
Primary Outcome 3 | 4 weeks
  Change in score in each group on Stait and Trait anxiety inventory (STAI)

SECONDARY OUTCOMES:
Secondary Score | 4 weeks
  Change in score on Self efficacy in Food Allergy Questionnaire (SEFAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Crealey, MD, Principal Investigator — Children's Health Ireland
Locations (1):
- Children's Health Ireland, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No